CLINICAL TRIAL: NCT00954603
Title: Compare Efficacy and Safety Between Quetiapine and Haloperidol in Treatment Delirium
Brief Title: A Double-blind, Randomized, Controlled Trial of Quetiapine Versus Haloperidol for the Treatment of Delirium
Acronym: QHdelirium
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: few delirious patients were enrolled.
Sponsor: Chiang Mai University (Other)
Responsible Party: Associate prof. Benchalak Maneeton, department of psychiatry, faculty of medicine, Chiang mai university, Thailand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MedCMU Que vs Halo - 2008; Que vs Halo - 2008 (Other: 077/2552)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-08

CONDITIONS: Delirium
Keywords: delirium rating scale; clinical global improvement; extrapyramidal side effect
MeSH Terms: conditions — Delirium | interventions — Quetiapine Fumarate; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- quetiapine (Experimental): atypical antipsychotic drug
  Interventions: Drug: quetiapine
- haloperidol (Active Comparator): typical antipsychotic drug
  Interventions: Drug: haloperidol

INTERVENTIONS:
Drug: quetiapine — 25-100 mg
  Other Names: seroquel
  Arms: quetiapine
Drug: haloperidol — 0.5-2 mg
  Other Names: haldol
  Arms: haloperidol

SUMMARY:
The purpose of this study is to determine whether quetiapine, and haloperidol are effective and safe in the treatment psychiatric symptoms in patients with delirium.

DETAILED DESCRIPTION:
A delirious state often founds in general hospitals and remains a significant cause of death. Existing methods of treatment includes identification and elimination of factors contributing to the delirium in addition to pharmacological and nonpharmacological treatment interventions (Trzepacz et al., 1999). Antipsychotics can play an important role in the management of the symptoms of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 -75 years
* Was admitted in Maharaj Nakhon Chiang Mai hospital
* Was diagnosed by the diagnostic criteria for DSM-IV-TR delirium due to a general medical condition or delirium due to multiple etiologies
* Delirious state (delirium) of the patients was confirmed by using name-assess confusion assessment method (CAM) and assessment of severity with delirium rating scale-revised-98 (DRS-R-98)
* Have a written consent from the legal representatives

Exclusion Criteria:

* Was diagnosed substance withdrawal delirium
* Having a history drug allergy either from quetiapine or haloperidol
* Female patients who are pregnant or breastfeeding
* No written consent from the legal representatives
* Received other anti-psychotic drug before attend the study
* Being ill with renal or hepatic failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
decrease in delirium rating scale and clinical global improvement | 7 days

SECONDARY OUTCOMES:
compare extrapyramidal and other report side effects of quetiapine and haloperidol from modified Simpson Angus scale and other report side effects. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Benchalak Maneeton, Assoc Prof, Principal Investigator — Department of Psychiatry,Faculty of Medicine, Chiang Mai university, Thailand
Locations (1):
- Department of psychiatry, faculty of medicine, Chiang Mai university, Chiang Mai, Thailand

REFERENCES:
- [Result] Maneeton B, Maneeton N, Srisurapanont M. An open-label study of quetiapine for delirium. J Med Assoc Thai. 2007 Oct;90(10):2158-63. PMID 18041437
- [Derived] Maneeton B, Maneeton N, Srisurapanont M, Chittawatanarat K. Quetiapine versus haloperidol in the treatment of delirium: a double-blind, randomized, controlled trial. Drug Des Devel Ther. 2013 Jul 24;7:657-67. doi: 10.2147/DDDT.S45575. Print 2013. PMID 23926422
- See also: treatment delirium — http://emedicine.medscape.com/article/288890-treatment
- See also: treatment delirium — http://www.icudelirium.org/
- See also: treatment delirium — http://en.wikipedia.org/wiki/Delirium#Treatment